CLINICAL TRIAL: NCT01739413
Title: Effect of Epidural Anesthesia and Analgesia on Insulin Secretion in Patients With Preoperative Decreased Insulin Sensitivity
Brief Title: Effect of Anesthesia on Insulin Secretion in Patients With Preoperative Decreased Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriele Baldini, MD, MSc, Assistant Professor (Other)
Responsible Party: Sponsor-Investigator, Gabriele Baldini, MD, MSc, Assistant Professor, Assitant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-263-SDR
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Anesthesia (Active Comparator): Patients will receive general anesthesia alone followed by intravenous morphine for postoperative pain control. This techniques is safe and is standard procedure for colorectal surgery.
  Interventions: Procedure: Anesthesia
- Epidural Anesthesia (Experimental): Patients will receive general anesthesia plus epidural anesthesia followed by epidural analgesia for postoperative pain control. This techniques is safe and standard procedure for colorectal surgery.
  Interventions: Procedure: Anesthesia

INTERVENTIONS:
Procedure: Anesthesia — Patients will be randomized to receive either epidural or general anesthesia for pain management throughout their surgery.

SUMMARY:
Epidural anesthesia has been found to manipulate the hyperglycemic response to surgery. It is unclear, however, whether the preoperative metabolic status of the surgical patient plays a role in the degree of this hyperglycemic response. For instance, the presence of low insulin sensitivity before surgery could predispose the individual to an altered metabolic response after surgery. In this case, it would be appropriate to identify adequate interventions that attenuate the response to surgical stress and facilitate the recovery process.

The aims of this research projects are the following:

1. To determine the extent in which epidural local anesthetics, initiated before surgery and continued after surgery, improves insulin secretion in patients with preoperative low insulin sensitivity.
2. To understand which measures of postoperative recovery are sensitive to the restoration of insulin secretion in this particular group of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving elective resection of malignant, non metastatic, colorectal lesions

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) health status class 4-5
* Dementia,neuromuscular disease, psychosis
* Cardiac abnormalities
* Severe end-organ disease such as cardiac failure (New York Heart Association classes I-IV)
* Chronic obstructive pulmonary disease
* Renal failure (creatinine > 1.5 mg/dl)
* Hepatic failure (liver transaminases >50% over the normal range)
* Diabetics with glycosylated hemoglobin > 6%
* Steroid consumption longer than 30 days sepsis
* Morbid obesity (body mass index >40)
* Anemia (hematocrit < 30 %, haemoglobin <10g/dl, albumin < 25mg/dl).
* Patients will be excluded if they have poor English or French comprehension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Hyperinsulinemic-euglycemic clamp | up to 2 days after surgery
  The Hyperinsulinemic-euglycemic clamp is the gold standard for measuring insulin sensitivity. Patients receive a 2 hour infusion of glucose and insulin, which is adjusted throughout the study period in order to maintain a blood glucose concentration at 5.5mmol/L. The test will take place one week before surgery and on the second postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Donatelli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Donatelli F, Corbella D, Di Nicola M, Carli F, Lorini L, Fumagalli R, Biolo G. Preoperative insulin resistance and the impact of feeding on postoperative protein balance: a stable isotope study. J Clin Endocrinol Metab. 2011 Nov;96(11):E1789-97. doi: 10.1210/jc.2011-0549. Epub 2011 Aug 31. PMID 21880795